CLINICAL TRIAL: NCT05308212
Title: Multicenter, Double-blind, Comparative, Randomized Tolerability, Safety and Immunogenicity Trial of the FLU-M® Tetra Inactivated Vaccine in Volunteers Aged 60 Years and Above
Brief Title: Tolerability, Safety and Immunogenicity Trial of the FLU-M® Tetra
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FLM-TE-04-2020
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: influenza; flu; vaccine; FLU-M Tetra
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FLU-M Tetra w/p (Experimental): 211 volunteers aged 60 y.o. and older received a single intramuscular dose of the Flu-M Tetra vaccine (with preservative) intramuscularly
  Interventions: Biological: Flu-M Tetra [Inactivated split influenza vaccine] w/p
- FLU-M Tetra w/o/p (Experimental): 211 volunteers aged 60 y.o. and older received a single intramuscular dose of the Flu-M Tetra vaccine (without preservative) intramuscularly.
  Interventions: Biological: Flu-M Tetra [Inactivated split influenza vaccine] w/o/p
- Ultrix (Active Comparator): 211 volunteers aged 60 y.o. and older received a single intramuscular dose of the Ultrix vaccine.
  Interventions: Biological: Ultrix [Inactivated split influenza vaccine]

INTERVENTIONS:
Biological: Flu-M Tetra [Inactivated split influenza vaccine] w/p — solution for intramuscular injection, 0.5 ml
  Arms: FLU-M Tetra w/p
Biological: Flu-M Tetra [Inactivated split influenza vaccine] w/o/p — solution for intramuscular injection, 0.5 ml
  Arms: FLU-M Tetra w/o/p
Biological: Ultrix [Inactivated split influenza vaccine] — solution for intramuscular injection, 0.5 ml
  Arms: Ultrix

SUMMARY:
Comparative assessment of the tolerability, safety, and immunogenicity of the FLU-M® Tetra quadrivalent inactivated split influenza vaccine and the Ultrix® vaccine in volunteers aged 60 years and above.

DETAILED DESCRIPTION:
Evaluation of the tolerability, safety and immunogenicity of the inactivated split influenza vaccine FLU-M® Tetra compared to Ultrix® vaccine in volunteers aged 60 years and above.

Volunteers were screened and randomized in three groups: the Flu-M Tetra w/p (with preservative) group, the Flu-M Tetra w/o/p (without preservative) group and the Ultrix® group. All subjects were followed up for 28 days post randomization and vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers (men and women) at the age of 60 years and above
2. Written informed consent of volunteers to participate in the clinical trial;
3. Volunteers able to fulfill requirements of the Protocol (i.e. fill out the patient's diary, come to follow-up visits);
4. For fertile women - a negative result of the pregnancy test and consent to observe adequate methods of contraception during the trial and at least two months after vaccination;
5. For fertile men - consent to observe adequate methods of contraception during the trial and at least two months after vaccination, except for men after vasectomy with documented azoospermia, and their sexual partners should use methods of contraception that ensure more than 90% reliability or be incapable of conception after a surgical sterilization or have a natural menopause for at least 2 years.

Exclusion Criteria:

1. History of influenza/ARVI or previous influenza vaccination during 6 months before the trial;
2. Positive result of the SARS-CoV-2 test;
3. A serious post-vaccination reaction (temperature above 40 °C, hyperemia or edema more than 8 cm in diameter) or complications (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions accompanied or not accompanied by a fever due to any previous vaccination);
4. Allergic reactions to vaccine components or any previous vaccination;
5. History of allergic reaction to chicken protein;
6. History of Guillain-Barré syndrome (acute polyneuropathy);
7. Previous vaccination with rabies vaccines less than 2 months before immunization or scheduled vaccination with rabies vaccines within 1 month after immunization with the trial vaccines;
8. History of leukemia, cancer, autoimmune diseases;
9. Positive blood test results for HIV, syphilis, hepatitis B/C.
10. Volunteers who received immunoglobulin or blood products or had a blood transfusion during the last three months before the trial;
11. History of long-term use (more than 14 days) of immunosuppressants or immunomodulatory drugs for six months before the trial;
12. History of any confirmed or suspected immunosuppressive or immunodeficiency condition;
13. History of chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, the gastrointestinal tract, liver, kidneys, hematopoietic, immune and endocrine system, mental disease in the acute stage or in the decompensation stage (recovery less than 4 weeks before vaccination);
14. History of eczema;
15. Treatment with glucocorticosteroids, including in small doses, as well as local use of drugs containing steroids (> 10 mg of prednisolone or its equivalent for more than 14 days before the screening);
16. Tuberculosis, neurological or mental disorders, a convulsive syndrome, including in the past medical history;
17. History of acute infectious diseases (recovery less than 4 weeks before vaccination);
18. Consumption of more than 10 units of alcohol per week or history of alcohol addiction, drug addiction or abuse of pharmaceutical products;
19. Smoking of more than 10 cigarettes per day;
20. Participation in another clinical trial during the last 3 months;
21. Pregnancy or lactation;
22. Coagulopathy, haemophilia;
23. Taking aspirin or other antiplatelet agents in high doses.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 633 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) ratio of antibodies after vaccination | days 0, 28
  Geometric mean titer (GMT) of antibodies in the blood serums of vaccinated people in haemagglutination inhibition assay.

SECONDARY OUTCOMES:
Change from baseline seroconversion rate at 28 days | days 0, 28
  Seroconversion rate refers to the percentage of subjects who have a prevaccination titer of influenza haemagglutinin antibody titer (HA titer) ≤ 1:10 and a post-vaccination HA titer ≥ 1:40 or a prevaccination HA titer > 1:10 and at least a 4-fold increase in post-vaccination HA titer vs. the baseline.
Seroconversion factor | days 0, 28
  Seroconversion factor is an increase in the geometric mean titers of antibodies at Day 28 vs. the baseline level, expressed in the fold rise.
Seroprotection rate | days 0, 28
  Seroprotection rate refers to the percentage of subjects with a generated protective HA titer (at least 1:40) vs. the baseline level.
Frequency of development of AEs associated with the vaccination | days 0-28
  An adverse event (AE) is any adverse medical occurrence in a trial subject who has received a pharmaceutical product or medicine that does not necessarily have a causal relationship with the medicine.
  AE include: new disease, complication of signs or symptoms of the condition being treated or a concomitant disease, effect of the trial drug or the reference drug, effect associated with a trial procedure, any combination of one or more of these factors.
Frequency of development of SAEs associated with the vaccination | days 0-28
  An adverse event is considered serious if it is fatal, threatens the life, requires hospitalization or extension of hospitalization, results in permanent or significant disability, is a congenital abnormality or defect (not applicable to this trial), is an important medical event.
Number of participants with abnormal physical examination findings | days 0,1,3,7,28
  Physical examination of volunteers includes an interview, discovery of complaints and symptoms, when required, palpation, auscultation, percussion for the following organs and systems: skin, mucosa, eyes, oral cavity and pharynx, lungs/chest, cardiovascular system, abdominal organs, nervous system, lymph nodes, musculoskeletal system, endocrine system.
Results of assessment of blood pressure (BP) | days 0,1,3,7,28
  BP measurements include the systolic and diastolic blood pressure.
Results of assessment of heart rate (HR) | days 0,1,3,7,28
  HR is measured during auscultation of the heart in parallel with determining the pulse rate on the radial artery (or on the carotid artery in case of weak pulsation in the radial artery) for a minute while sitting.
Results of E immunoglobulin tests | days 0,3,28
  Determination of total IgE.
Results of assessment of respiratory rate (RR) | days 0,1,3,7,28
  RR is measured for a minute at rest in the sitting position, by registering the breathing movements of the chest or abdominal wall, without attracting the patient's attention.
Results of assessment of body temperature | days 0,1,3,7,28
  Body temperature is measured with a mercury or digital thermometer in the armpit for at least 5 minutes or with a non-contact infrared digital thermometer.
Number of participants with abnormal neurological examinations | days 0,1,3,7,28
  Assessement of neurological status, cranial nerve function, motor sphere, reflex sphere, sensitive sphere, coordination sphere, pelvic functions, higher mental functions.
Number of participants with abnormal ECG findings | days 0,3
  ECG QT Interval, QTc Interval, PQ Interval, QRS complex.
Number of participants with abnormal complete blood counts results | days 0,3
  Hemoglobin, hematocrit, erythrocytes, leukocytes, platelets, leukocyte count, ESR.
Number of participants with abnormal biochemical blood tests results | days 0,3
  Total protein, creatinine, urea, glucose, total bilirubin, total cholesterol, AST, ALT, ALP.
Number of participants with abnormal urinalysis results | days 0,3
  pH, specific gravity, protein, glucose, red blood cells, white blood cells

CONTACTS AND LOCATIONS:
Locations (11):
- Russia (11):
  - State Autonomous Health Institution "Engels City Clinical Hospital No1", Engel's
  - Limited Liability Company Professorskaya Clinica, Perm
  - Limited Liability Company Energia Zdorovya, Saint Petersburg
  - Limited Liability Company MEDICINSKAYA CLINIKA, Saint Petersburg
  - Limited Liability Company Scientific Research Center Eco-Bezopasnost, Saint Petersburg
  - Piramida Limited Liability Company, Saint Petersburg
  - Private Health Care Institution Clinical Hospital "RZD-Medicine" in Saint Petersburg, Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "State Polyclinic No. 117", Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "State Polyclinic No. 43", Saint Petersburg
  - Limited Liability Company "DNA Research Center", Saratov
  - Federal State Budget Healthcare Institution "Yaroslavl Region Clinical Hospital No. 2", Yaroslavl